CLINICAL TRIAL: NCT04366674
Title: The Possible Effect of Modified Restoration of Tensor Veli Palatini on Audiological and Otological Outcome in Cleft Palate Repair.
Brief Title: Mordified Restoration of Tensor Veli Palatini in Cleft Palate Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lian Zhou, Prof., Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-K1145
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Langerbeck's repair (Active Comparator): Langerbeck's repair of cleft palate,without specific restoration of levator veli palatini or tensor veli palatini. Incisions along the margins of the cleft at the junction of oral and nasal mucosa. Lateral relaxing incisions were performed and the mucoperiosteal flap of hard palate were elevated on both sides except the ones with only soft palate cleft. The anterior end of the mucoperiosteal flap may be cut off for the purpose of tension relieving and would be resutured to the anterior area during closing. In the soft palate, the division was made between the oral mucous layer and the palatal musculature layer. Hamulus were broken for closing the cleft without tension. Closing was done by two seperated layers, one layer of nasal mucosa-palatal muscle, and one layer of oral mucosa.
  Interventions: Procedure: cleft palate repair
- restoration of levator veli palatini (Active Comparator): The incision was made similar to Langerbeck's repair. During disection, the levator veli palatini was identified after the elevation of flap. The levator veli palatini was separate from the oral and nasal mucosa. During closing, the anterior end of levator veli palatini was rotated towards the midline and the two muscle bundle from the two sides were sutured in the midline. In this process, the tensor veli palatini was not intentionally identified or dissected.
  Interventions: Procedure: cleft palate repair
- mordified restoration of tensor veli palatini (Experimental): Incision was made similar to Langerbeck's repair. During disection, the tensor veli palatini was identified after flap elevation. Its tendinous fibers was released from but still connected to the pterygoid process without breaking the hamulus or cutting off the tendinous fibers. If the tension is too strong during suturing, the tensor tendon could be partly dissected laterally meanwhile be kept continuity medially so that the tensor veli palatini could be rotated more medially. The levator veli palatini, tensor veli palatini, together with the palatine aponeurosis and the nasal mucosa from two sides were sutured in the middle line. The tensor veli palatini may not be jointed to the contralateral one directly.
  Interventions: Procedure: cleft palate repair

INTERVENTIONS:
Procedure: cleft palate repair — restoration of tensor veli palatini for the purpose of the muscle function recovery.

SUMMARY:
to study the benefical audiological and/or otological effect by mordified restoration of tensor veli palatini in cleft palate repair compared to traditional Langenbeck's repair and merely levator veli palatini restoration.

DETAILED DESCRIPTION:
71 patients with cleft palate received surgery were divided into 3 groups. Group 1: patients who received Langenbeck surgery without specific restoration of levator veli palatini or tensor veli palatini. Group 2: patients who received palate surgery with special levator veli palatini restoration. Group 3: patients who received palate surgery with modified tensor veli palatini restoration. The conductive auditory brainstem response and 226 Hz tympanometry were used to test the audiological and otological status of the three groups. Preoperative and postoperative results were compared intragroup and intergroup.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cleft palate.
* Primary palate repair.

Exclusion Criteria:

* Severe general disease
* Confirmed hereditary hearing loss or neuropathic hearing loss.
* Received any kind of audiological or otological therapy before.
* Patients and/or his/her don't want to continue the clinical trial.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Hearing level | 3 months after surgery
  Auditory brainstem response was tested in all three groups after surgery. The air conductive hearing threshold was used to assess the hearing level.
The otological status of middle ear | 3 months after surgery
  226 tympanometry was tested in all three groups after surgery. The results of 226 Hz tympanometry were classified based on Liden/Jerger classification. Four classes of tympanometry results were included.
Hearing level | 0 to 3 months before surgery
  Auditory brainstem response was tested in all three groups before surgery. The air conductive hearing threshold was used to assess the hearing level.
The otological status of middle ear | 0 to 3 months before surgery
  226 tympanometry was tested in all three groups before surgery. The results of 226 Hz tympanometry were classified based on Liden/Jerger classification. Four classes of tympanometry results were included.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Zhou, D.D.S, Principal Investigator — Peking Union Medical College Hospital